CLINICAL TRIAL: NCT07206680
Title: Effect of Extracorporeal Shockwave Therapy on Pruritus in Neurodermatitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abd Al Rahman Khaled Muhammed Muhammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005978
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Neurodermatitis
MeSH Terms: conditions — Neurodermatitis | interventions — Extracorporeal Shockwave Therapy; Emollients; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave therapy + corticosteroids + emollients (Experimental): It will include 17 patients suffering from neurodermatitis who will receive shockwave therapy for 10min, 4 sessions, once per week and emollients & corticosteroids for a month.
  Interventions: Device: Shockwave therapy; Drug: Emollients & corticosteroids
- Corticosteroids & Emollients (Active Comparator): It will include 17 patients suffering from neurodermatitis who will receive their emollients & corticosteroids only for a month.
  Interventions: Drug: Emollients & corticosteroids

INTERVENTIONS:
Device: Shockwave therapy — The procedures for Extracorporeal Shockwave Therapy (ESWT) involve several steps. First, the patient is positioned comfortably, and the physiotherapist explains the treatment procedure. Before the session begins, the device cables are checked for proper functioning. The shockwave type used is Non-Focused/Radial, with a treatment duration not exceeding 10 minutes. The frequency is set at 4 Hz, and the intensity ranges from 0.05 to 0.20 mJ/mm². Each session involves a total of 1000 to 2000 shocks. The treatment consists of four sessions, each held once a week.
  Arms: Shockwave therapy + corticosteroids + emollients
Drug: Emollients & corticosteroids — Patients in both groups will receive emollients & corticosteroids for one month.

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect of shockwave therapy on reducing pruritus in neurodermatitis patients.

DETAILED DESCRIPTION:
Based on the occurrence of side effects caused by conventional medication for prolonged employment, dermatologists and patients show solicitude for multifaceted effective methods to control the chronic and relapsing nature of neurodermatitis.

Although new modalities are continuously coming up for pruritus, there remains a great gap for providing symptom relief.

Furthermore, there is a lack in the quantitative knowledge and information in the published studies about benefits of shockwave therapy on the treatment of pruritus in neurodermatitis patients. So, this study is designed to outline the therapeutic efficacy of shockwave therapy on the treatment of pruritus in neurodermatitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 55:75 years.
* Male and female patients will participate in the study.
* All patients have neurodermatitis.
* All patients will be received the same approach of medication and nursing care.
* All patients enrolled in the study will have their informed consent.

Exclusion Criteria:

* Patients diagnosed with cancer.
* Pregnant woman.
* active infection.
* Patients with any systemic diseases that may interfere with the objectives of the study.
* Cardiac pacemakers or other implantable devices.
* Current anticoagulation use.
* Any other cause of itching

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
5-D Itching Scale | one month
  The 5-D Itching Scale will be used to assess the improvement of cases by evaluating pruritus severity. Patients will complete the scale both before starting the treatment and at four sessions following the treatment. The following steps will be followed during the assessment: the patient will be positioned comfortably (sitting position), the physiotherapist will explain the pruritus symptoms score to the patient, and the patient will determine their points on the 5-D itch scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nessrien Afify Abd El Rashid, PhD, Study Chair — Assistant Professor, Cairo University; Noha Zakaria Tawfik, PhD, Study Director — Assistant Professor, Suez Canal University; Doaa Atef Aly, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt